CLINICAL TRIAL: NCT03107559
Title: Can the Perfusion Index be Used as an Objective Instrument for the Assessment of Pain in the Labor Analgesia?
Brief Title: Perfusion Index and Labor Analgesia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Erzincan University (Other)
Responsible Party: Principal Investigator, ILKE KUPELI, assist. prof., Erzincan University
Other Study IDs: ERZINCAN UNIVERSITY pain&pi
Record Dates: First submitted 2017-04-05; First posted 2017-04-11 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: perfüsion Index in Removal of the Epidural Analgesia
Keywords: perfüsion index; epidural analgesia; labor

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: perfüsion index — Determination of the relationship between VAS values and PI in patients with normal delivery who undergo epidural analgesia

SUMMARY:
It can be suggested that sympathetic tonus increase and pain, caused by the removal of the effect of epidural analgesia applied at birth, may also affect perfüsion index. The purpose of this study is; To correlate the VAS value at the time of return of epidural analgesia with the PI values at that time and, to test the possibility of using PI variants as an objective tool for predicting pain initiation time and assessing pain.

ELIGIBILITY:
Inclusion Criteria:

* women who will give normal spontaneous vaginal delivery
* Between the ages of 18-45

Exclusion Criteria:

* Patients who do not accept the procedure,
* those under 18 years of age - over 45 years,
* those with low platelet counts,
* those with infection at the puncture site,
* those with progressive neurological disease,
* Those with increased intracranial pressure,
* those with hypovolemia

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: 30 women between the ages of 18-45 who will give normal spontaneous vaginal delivery
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-05-30 (Estimated); Primary Completion 2017-07-15 (Estimated); Study Completion 2017-08-01 (Estimated)

PRIMARY OUTCOMES:
relationship between Visual analogue scale and Perfüsion index | three month
  Determination of the relationship between VAS values and PI in patients with normal delivery who undergo epidural analgesia,

SECONDARY OUTCOMES:
relationship between heart rate and Perfüsion index | three month
  Determination of the relationship between heart rate and PI in patients with normal delivery who undergo epidural analgesia,
relationship between non-invazive blood pressure and Perfüsion index | three month
  Determination of the relationship between non-invazive blood pressure and PI in patients with normal delivery who undergo epidural analgesia,

CONTACTS AND LOCATIONS:
Overall Officials: ilke kupeli, Principal Investigator — Erzincan University
Locations (1):
- Erzincan University, Erzincan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Breivik H, Borchgrevink PC, Allen SM, Rosseland LA, Romundstad L, Hals EK, Kvarstein G, Stubhaug A. Assessment of pain. Br J Anaesth. 2008 Jul;101(1):17-24. doi: 10.1093/bja/aen103. Epub 2008 May 16. PMID 18487245
- [Background] Tousignant-Laflamme Y, Marchand S. Sex differences in cardiac and autonomic response to clinical and experimental pain in LBP patients. Eur J Pain. 2006 Oct;10(7):603-14. doi: 10.1016/j.ejpain.2005.09.003. Epub 2005 Nov 18. PMID 16298532
- [Result] Ledowski T, Ang B, Schmarbeck T, Rhodes J. Monitoring of sympathetic tone to assess postoperative pain: skin conductance vs surgical stress index. Anaesthesia. 2009 Jul;64(7):727-31. doi: 10.1111/j.1365-2044.2008.05834.x. Epub 2009 Jan 28. PMID 19183409
- [Result] Bird J. Selection of pain measurement tools. Nurs Stand. 2003 Dec 10-16;18(13):33-9. doi: 10.7748/ns2003.12.18.13.33.c3515. PMID 14694870
- [Result] Nishimura T, Nakae A, Shibata M, Mashimo T, Fujino Y. Age-related and sex-related changes in perfusion index in response to noxious electrical stimulation in healthy subjects. J Pain Res. 2014 Feb 10;7:91-7. doi: 10.2147/JPR.S57140. eCollection 2014. PMID 24550680